CLINICAL TRIAL: NCT06554249
Title: Full Bladder IUD Insertion Without Vulsellum Under Ultrasound Guidance Versus the Standard Technique for IUD Insertion
Brief Title: Full Bladder IUD Insertion Without Vulsellum Under Ultrasound Guidance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Bedaya Hospital (Other)
Responsible Party: Principal Investigator, Usama M Fouda, Prof., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUD/Ultrasound
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Contraceptive Device
Keywords: IUD; Ultrasound; Full bladder; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vulsellum group (Active Comparator): The patients are asked to empty the bladder before IUD insertion. The vulsellum is applied on the cervix, sounding of the uterus is done and the IUD is inserted according to the standard technique of IUD insertion.
  Pain intensity is assessed after the procedure using a visual analogue scale.
  Interventions: Procedure: Vulsellum group
- Ultrasound group (Active Comparator): During the two hour period before IUD insertion, the patients are asked to drink about one liter of water and to avoid micturition.
  Abdominal ultrasound is used to obtain a sagittal view of the uterus and the IUD is introduced into the uterine cavity under ultrasound guidance.
  The vulsellum and uterine sound are not used during IUD insertion. Pain intensity is assessed after the procedure using a visual analogue scale.
  Interventions: Procedure: Ultrasound group

INTERVENTIONS:
Procedure: Vulsellum group — The patients are asked to empty the bladder before IUD insertion. The vulsellum is applied on the cervix, sounding of the uterus is done and the IUD is inserted according to the standard technique of IUD insertion.
  Pain intensity is assessed after the procedure using a visual analogue scale.
  Arms: Vulsellum group
Procedure: Ultrasound group — During the two hour period before IUD insertion, the patients are asked to drink about one liter of water and to avoid micturition.
  Abdominal ultrasound is used to obtain a sagittal view of the uterus and the IUD is introduced into the uterine cavity under ultrasound guidance.
  The vulsellum and uterine sound are not used during IUD insertion. Pain intensity is assessed after the procedure using a visual analogue scale..
  Arms: Ultrasound group

SUMMARY:
The aim of this study is to determine whether full bladder IUD insertion without vulsellum or uterine sound under ultrasound guidance is associated with less pain compared with the standard technique of IUD insertion .

DETAILED DESCRIPTION:
The intrauterine device (IUD) is an effective method of contraception. Pain experienced during IUD insertion is one of the main causes that limits its widespread use.

Pain during IUD insertion is caused by insertion of cusco vaginal speculum, sounding the uterus, application of vulsellum to grasp the cervix, the passage of the inserter tube through the cervical canal and uterine cavity..

In order to minimize the pain associated with IUD insertion , several studies reported that the use of ultrasound to guide the insertion of IUD into uterine cavity was associated with less pain and more accurate placement of IUD, other studies reported that filling the bladder during IUD insertion minimized the pain associated with IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

* Women requesting IUD insertion

Exclusion Criteria:

* Active pelvic infection
* Viable intrauterine pregnancy
* Uterine anomalies
* Uterine fibroid
* Wilson disease

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | Immediately after the procedure
  Measured using 100 mm visual analogue scale ( 0 = no pain and 100 = worst possible pain)

SECONDARY OUTCOMES:
Success of IUD insertion | Immediately after the procedure
  ( number of successfully inserted IUD / total number of IUD insertion attempts)

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Prof., Principal Investigator — Cairo University
Locations (1):
- Faculty of medicine, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baradwan S, Alshahrani MS, Alnoury A, Khadawardi K, Khan MA, Abdelkader RAA, Saleh OI, Galal HM, Mohamed SMA, Abdelhakim AM, Elgedawy AM, Elbahie AM, Gaber MA, Magdy AA, Shaheen K. Does Ultrasound Guidance Provide Pain Relief During Intrauterine Contraceptive Device Insertion? A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Ultrasound Med. 2023 Jul;42(7):1401-1411. doi: 10.1002/jum.16166. Epub 2022 Dec 30. PMID 36583454